CLINICAL TRIAL: NCT05369715
Title: Diurnal Variation of the Effect of Aerobic Exercise on Glycemic Metabolism and Fat Oxidation in Humans: Role of Sex
Brief Title: Diurnal Variation of Exercise on Metabolic Health
Acronym: DIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Director, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DIVA project
Record Dates: First submitted 2021-12-24; First posted 2022-05-11 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Aerobic Exercise; Acute Exercise; Circadian Rhythm Sleep-Wake Disorders, Unspecified Type; Glucose Metabolism; Lipid Metabolism; Diurnal Variation; Young Adults
Keywords: Aerobic Exercise; Diurnal Variation; Circadian Rhythm; Glucose Metabolism; Lipid Metabolism; Young adults
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To blind this study is not possible due to the studied conditions: morning and evening. Only data assesors can be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning (Experimental): 60 minutes cycling on cycle ergometer in the morning (11:30). Steady-state test at an intensity of 65% of participant's heart rate reserve.
  Interventions: Other: Exercise
- Evening (Experimental): 60 minutes cycling on cycle ergometer in the evening (18:30). Steady-state test at an intensity of 65% of participant's heart rate reserve.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Aerobic exercise

SUMMARY:
The main objective of this project is to study the diurnal variation of the effect of exercise on glycemic metabolism and fat oxidation in humans.

DETAILED DESCRIPTION:
Strong scientific evidence supports the beneficial effects of exercise on cardiovascular health, the regulation of glucose metabolism, and fat oxidation. Physical performance capacity is known to fluctuate throughout the day, however, it is unknown whether there is an optimal time of day to maximize the effects of exercise on health, and specifically on blood glucose metabolism and fat oxidation. Finding the ideal time to perform physical exercise is of clinical and public health interest. Likewise, optimizing the timing of physical exercise to coincide with the greater physiological response of each individual would mean increasing the potential of exercise as a therapeutic tool.

Specific aims of this project are a) to describe possible differences dependent on sex in the diurnal variation of the effect of exercise on glycemic metabolism and fat oxidation, and b) to characterize the molecular mechanisms implicated.

18 men and 17 women with normal weight will be randomized into two conditions (morning and evening) with at least 3 days of separation in between. Each evaluation will conform the following tests:

1. Basal metabolic rate assessment through indirect calorimetry during 30 minutes.
2. Fuel oxidation and energy expenditure assesment during a 60 minutes bout of aerobic steady-state exercise (cycling), through indirect calorimetry.
3. Fuel oxidation and energy expenditure assesment after exercise during 30 minutes, through indirect calorimetry.
4. Blood samples assesment before, inmediately after, and 90 minutes after exercise.
5. Quadriceps biopsies before, and inmediately after exercise. *This will be done only in a sub-cohort.
6. Visual analog scales to assess appetite before, inmediately after, and 90 minutes after exercise.
7. Continous glucose monitoring from the previous 24 hrs to first session day, until 48 hrs after the last exercise session.

Previous to this, participants' body composition and fitness level will be assesed via densitometry and a maximal exercise test, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index: 18.5to 27.0 kg/m2.
* Physical activty < 5 days/week.
* To be able to understand instrucctions, objectives and study protocol.

Exclusion Criteria:

* History of a major adverse cardiovascular event, kidney failure, cirrhosis, eating disorder, weight control surgery, or HIV / AIDS.
* Rheumatoid arthritis, Parkinson's disease, active cancer treatment in the past year, type 1 diabetes mellitus, or another medical condition for which fasting is contraindicated.
* Any condition that, in the judgment of the investigator, impairs the ability to participate in the study or poses a personal risk to the participant.
* Use of medications that may affect the results of the study.
* Unstable body weight for 3 months before the start of the study (> 4 kg weight loss or gain)
* Pregnancy and breastfeeding.
* Active tobacco abuse or illicit drug use or a history of alcohol abuse treatment.
* On a special diet or prescribed for other reasons (eg celiac disease).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change from resting blood glucose to 48 hours after exercise | 4 days. Pre exercise day, exercise day, post-24hrs exercise day, post-48hrs exercise day.
  A continuous glucose monitor inserted into the skin of the arm upper forearm area will be used to record and store blood glucose levels every 15 minutes, for 24 hours, 14 consecutive days. Within this time range both exercise conditions will be performed. The monitor will be placed 24 hours before the first exercise session and will be removed 48 hours after the second exercise session. Therefore, change from resting blood glucose 24 hours previous to 48 hours after exercise will be obtained for each condition.
Change from resting fat oxidation to 90 minutes after exercise | 210 minutes
  Participants will lay down for 60 minutes where resting gas exchange was measured (using a canopy hood for gases collection) for 30 minutes in two separated 15 minutes stages, corresponding to 45 to 60 and 75 to 90 minutes after exercise, respectively
Change from resting markers of glucose metabolism to 90 minutes after exercise | 180 minutes
  Blood samples will be taken after exercise, immediately after exercise and 90 minutes after exercise, in order to measure change in plasma concentration of markers of glucose metabolism from resting to 90 minutes after exercise.
Change from resting markers of fatty acid metabolism to 90 minutes after exercise | 180 minutes
  Blood samples will be taken to measure plasma concentration of markers of fatty acid metabolism before, immediately after and 90 minutes after exercise.
Gene expression | 90 minutes
  Muscular biopsies will be taken from the vastus lateralis' distal part of the quadriceps in a sub-sample before and immediately after the exercise. Biopsies will be performed by an experienced surgeon using microbiopsy needles (Achieve Automatic Needle 16G x 15 cm), obtaining ~30 mg per biopsy after previous local anaesthesia with 2% lidocaine. From each time point (Pre and Post), 1 skeletal muscle samples will be collected and immersed in liquid nitrogen and stored at -80ºC until further analysis (i.e.: transcriptomics). RNA from skeletal muscle will be extracted using Trizol (Invitrogen).
Protein expression | 90 minutes
  Muscular biopsies will be taken from the vastus lateralis' distal part of the quadriceps in a sub-sample before and immediately after the exercise. Biopsies will be performed by an experienced surgeon using microbiopsy needles (Achieve Automatic Needle 16G x 15 cm), obtaining ~30 mg per biopsy after previous local anaesthesia with 2% lidocaine. From each time point (Pre and Post), 1 skeletal muscle samples will be collected and immersed in liquid nitrogen and stored at -80ºC until further analysis (i.e.: proteomics).
Mitochondrial breathing | 90 minutes
  Muscular biopsies will be taken from the vastus lateralis' distal part of the quadriceps in a sub-sample before and immediately after the exercise. Biopsies will be performed by an experienced surgeon using microbiopsy needles (Achieve Automatic Needle 16G x 15 cm), obtaining ~30 mg per biopsy after previous local anaesthesia with 2% lidocaine. From each time point (Pre and Post), 1 skeletal muscle samples will be collected and treated fresh to study mitochondrial respiration.
Mitochondrial supercomplexes | 90 minutes
  Muscular biopsies will be taken from the vastus lateralis' distal part of the quadriceps in a sub-sample before and immediately after the exercise. Biopsies will be performed by an experienced surgeon using microbiopsy needles (Achieve Automatic Needle 16G x 15 cm), obtaining ~30 mg per biopsy after previous local anaesthesia with 2% lidocaine. From each time point (Pre and Post), 1 skeletal muscle samples will be collected and immersed in liquid nitrogen and stored at -80ºC until further analysis (i.e.: mitochondrial protein supercomplexes by blue-native PAGE).

SECONDARY OUTCOMES:
Change from resting appetite to 90 minutes after exercise | 180 minutes
  Measures of appetite before, immediately after and 90 minutes after exercise using an appetite visual analog scale (appetite VAS) scoring from 0 to 10, where 0 is the minimum punctuation for appetite and 10 is the maximum punctuation for appetite.

OTHER OUTCOMES:
Continous body temperature | 255
  Before, during and after exercise, periodic recordings of the central and distal temperature will also be made by using thermal iButtons (iButtons DS 1922 L, Maxim, Dallas, USA).
Diet | 4 days. Pre-exercise day, exercise day, post-24 hrs exercise and post-48 hrs exercise
  Standarditation and control of diet. Diet will be standardized 24 hours prior to each exercise session (55% carbohydrates, 27% fat and 18% proteins). In addition, diet will be monitored for 48 hours after the exercise test.
Physical activity | 4 days. Pre-exercise day, exercise day, post-24 hrs exercise and post-48 hrs exercise
  Levels of physical activity will be controlled by accelerometry 24 hours before and 48 hours after each exercise session (Actigraph, GT3X).
Body composition | 7 minutes
  Body fat percentage will be evaluated by dual X-ray absorptiometry (Discovery Wi, Hologic, Inc, Bedford, MA, USA).
Body mass index (BMI) | 5 minutes
  Weight and height will be measured (Seca model 799, Electronic Column Scale, Hamburg, Germany). Weight and height measurements will be aggregated to obtain BMI in kg/m^2
Chronotype | 15 minutes
  Participants will complete the HÖME questionnaire, that determines chronotype (morning-evening).
Menstrual cycle | 5 minutes
  Dates of the different phases of the menstrual cycle will be recorded in order to locate all tests in the luteal phase. However, we have observed that fat oxidation is not affected by the phase of the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Ruiz Ruiz, Dr., Principal Investigator — Granada University
Locations (1):
- University of Granada - Instituto Mixto Universitario Deporte y Salud, Granada, Spain